CLINICAL TRIAL: NCT03573882
Title: An Open Label Extension Study of Voxelotor (GBT440) Administered Orally to Participants With Sickle Cell Disease Who Have Participated in Voxelotor Clinical Trials
Brief Title: Study to Assess the Effect of Long-term Treatment With Voxelotor in Participants Who Have Completed Treatment in Study GBT440-031
Acronym: 034OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Emerging clinical data evaluated by Pfizer and shared with regulatory authorities indicates that the risk profile of voxelotor in people with SCD exceeds the benefits observed in previously generated global research and requires further assessment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBT440-034; C5341022 (Other: Alias Study Number)
Expanded Access: NCT03943615 (No longer available)
Record Dates: First submitted 2018-05-15; First posted 2018-06-29 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: Open Label Extension
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Voxelotor (Other): Participants will receive voxelotor (GBT440) at the highest dose (either 900 mg or 1500 mg) deemed safe by the Data Safety Monitoring Board (DSMB).
  Interventions: Drug: Voxelotor

INTERVENTIONS:
Drug: Voxelotor — 300mg or 500mg Tablet, Oral, With or Without Food
  Other Names: GBT440

SUMMARY:
Open Label Extension Study of Voxelotor Clinical Trial Participants with Sickle Cell Disease Who Participated in Voxelotor Clinical Trials

DETAILED DESCRIPTION:
This open label extension (OLE), multi-center study will be conducted at approximately 100 clinical sites globally and will be available to eligible participants from study GBT440-031.

The study will enroll participants from GBT440-031 (approximately 435) under any of the following conditions:

* Participant has completed 72 weeks of treatment regardless of dose selection for GBT440-031
* Dose selection has occurred for GBT440-031 and participant is on non-selected dose on GBT440-031
* GBT440-031 study interim data analysis and/or study modifications have occurred
* GBT440-031 study has completed

The objective of this open-label extension (OLE) study is to assess the long-term safety and treatment effect of voxelotor in participants who have completed treatment in study GBT440-031, using the following parameters:

1. Safety based upon AEs, clinical laboratory tests, physical examinations (PE) and other clinical measures.
2. Frequency of sickle cell disease (SCD)-related complications.
3. Hemolytic anemia as measured by hematological laboratory parameters (e.g. hemoglobin, reticulocytes and unconjugated bilirubin).

All participants will receive daily voxelotor treatment.

Participants may receive study drug as long they continue to receive clinical benefit which outweighs risk as determined by the Investigator and/or until the participant has access to voxelotor from an alternative source (i.e., commercialization or through a managed access program).

ELIGIBILITY:
Inclusion Criteria:

* Male or female study participants with SCD who participated and received study treatment in Study GBT440-031.

Note: Participants in GBT440-031 who discontinued study drug due to an AE, but who remained on study may be eligible for treatment in this study provided the AE does not pose a risk for treatment with voxelotor.

* Females of child-bearing potential are required to have a negative urine pregnancy test prior to dosing on Day 1.
* Female participants of child-bearing potential must use highly effective methods of contraception to 30 days after the last dose of study drug. Male participants must use barrier methods of contraception to 30 days after the last dose of study drug.
* Participant has provided written informed consent or assent (the ICF must be reviewed and signed by each participant; in the case of pediatric participants, both the consent of the participant's legal representative or legal guardian, and the participant's assent must be obtained).

Exclusion Criteria:

* Female who is breast-feeding or pregnant.
* Participant withdrew consent from Study GBT440-031.
* Participant was lost to follow-up from Study GBT440-031.
* Participant requiring chronic dialysis.
* Any medical, psychological, safety, or behavioral conditions, which, in the opinion of the Investigator, may confound safety interpretation, interfere with compliance, or preclude informed consent.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (34):
  - Arkansas Primary Care Clinic, PA, Little Rock, Arkansas
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Jackson Memorial Hospital (Investigational Drug Services), Miami, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Hospital & Clinics/SCCC, Research Pharmacy (Investigational Drug Services), Miami, Florida
  - University of Miami, Miami, Florida
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois Hospital and Health Science System, Chicago, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - St. Jude Affiliate Clinic Baton Rouge, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group-Medical Oncology, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sickle Cell Infusion Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital Research Pharmacy, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Montefiore - Einstein Center for Cancer Care, The Bronx, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Drug Service, Duke University Hospital, Durham, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Comprehensive Sickle Cell Clinic, Charleston, South Carolina
  - Medical University of South Carolina: Investigational Drug Services Pharmacy, Charleston, South Carolina
  - Methodist Comprehensive Sickle Cell Clinic, Memphis, Tennessee
  - Texas Children's Hospital - Investigational Pharmacy, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Clinical Research Services Unit- Virginia Commonwealth University, Richmond, Virginia
- Toronto General Hospital-University Health Network, Toronto, Ontario, Canada
- Egypt (6):
  - Alexandria Clinical Research Center, Faculty of Medicine, Alexandria University, Alexandria
  - Alexandria Clinical Research Center, Faculty of Medicine, Alexandria
  - Zagazig University Hospital, Alsharkia
  - Abu El Rich Hospital,Cairo University Hospital, Cairo
  - Ain Shams University Hospital, Cairo
  - The Egyptian Thalassemia Association ( E.T.A), Cairo
- Hôpital Européen Georges Pompidou - Medecine Interne, Paris, France
- Azienda Ospedaliera di Padova, Padua, Padova Veneto, Italy
- Kenya (3):
  - Centres for Disease Control and Prevention, Siaya, Kisumu County
  - KEMRI/CRDR - Kenya Medical Research Insititute - Center for respiratory Disease Research, Nairobi
  - Gertrude's Children's Hospital, Nairobi
- Lebanon (2):
  - American University of Beirut, Beirut
  - Nini Hospital, Tripoli
- Netherlands (2):
  - Academic Medical Center(AMC), Amsterdam
  - ErasmusMC, Rotterdam
- Sultan Qaboos University Hospital, Muscat, Oman
- Turkey (Türkiye) (3):
  - Adana Acibadem Hospital, Adana
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Mersin Universitesi Tip Fakultesi Saglik Arastirma ve Uygulama Hastanesi, Mersin
- United Kingdom (6):
  - Barts Health NHS Trust, London, Greater London
  - Homerton University Hospital NHS Foundation Trust, London, Greater London
  - Guys and St. Thomas Hospital NHS Foundation Trust, Great Maze Pond, London
  - King's College Hospital, London
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - McMillan Cancer Centre, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT440-034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label extension (OLE) study which included eligible participants from study GBT440-031 (NCT03036813). All participants were administered voxelotor 1500 milligrams (mg) in this study. Results were stratified according to previous treatment in GBT440-031 (NCT03036813).
Pre-assignment Details: A total of 179 participants were enrolled in the study. The study was terminated as emerging clinical data observed in studies other than the current study (GBT440-034) indicated that risk profile of voxelotor in people with sickle cell disease (SCD) exceeded benefits observed in previously generated global research and required further assessment.
Groups:
- Prior Treatment of Placebo in GBT440-031 (NCT03036813): Participants who received placebo in study GBT440-031 (NCT03036813) were administered voxelotor 1500 mg once daily in this study as long as they received clinical benefit and/or until the participant had access to voxelotor from an alternative source.
- Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813): Participants who received voxelotor 900 mg in study GBT440-031 (NCT03036813) were administered voxelotor 1500 mg once daily in this study as long as they received clinical benefit and/or until the participant had access to voxelotor from an alternative source.
- Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813): Participants who received voxelotor 1500 mg in study GBT440-031 (NCT03036813) were administered voxelotor 1500 mg once daily in this study as long as they received clinical benefit and/or until the participant had access to voxelotor from an alternative source.
Period: Overall Study
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813)
Started | 63 | 58 | 58
Treated | 62 | 58 | 58
Completed | 16 | 11 | 19
Not Completed | 47 | 47 | 39
Not completed — Study Terminated by Sponsor | 22 | 17 | 18
Not completed — Withdrawal by Subject | 6 | 11 | 7
Not completed — Adverse Event | 7 | 5 | 6
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Physician Decision | 4 | 3 | 2
Not completed — Participant is Noncompliant with Study Drug | 1 | 2 | 1
Not completed — Pregnancy | 1 | 2 | 0
Not completed — Other | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received treatment with study drug voxelotor in current study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813) | Total
Number analyzed (Participants) | 62 | 58 | 58 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.5 (10.80) | 28.5 (11.90) | 29.0 (13.00) | 28.7 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 37 | 100
  Male | 34 | 23 | 21 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 1 | 9
  Not Hispanic or Latino | 57 | 55 | 56 | 168
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 14 | 8 | 12 | 34
  Arab | 9 | 10 | 9 | 28
  Asian | 0 | 0 | 1 | 1
  Black or African American | 26 | 27 | 26 | 79
  Middle Eastern | 5 | 2 | 2 | 9
  White | 4 | 5 | 4 | 13
  Other | 2 | 2 | 0 | 4
  Multiple | 2 | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sickle Cell Disease (SCD)-Related Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs were defined as AEs with onset on or after the date of informed consent until 28 days after last dose of study drug. SCD-related TEAEs included preferred terms (PTs) of sickle cell anaemia with crisis, acute chest syndrome (ACS), pneumonia, priapism, and osteonecrosis. The number of participants with any SCD-related TEAEs was reported in this outcome measure.
Time Frame: From date of informed consent up to 28 days after last dose of study drug (maximum up to 300.7 weeks)
Population: The safety population included all enrolled participants who received treatment with study drug voxelotor in the current study.
Measure: Count of Participants; unit: Participants
Groups:
- Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813): Participants who received voxelotor 1500 mg in study GBT440-031 (NCT03036813) were administered voxelotor 1500 mg once daily in this study as long as they received clinical benefit and/or until the participant had access to voxelotor from an alternative source.
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
Participants | 47 | 42 | 42

2. Primary Outcome: Number of Participants With Non- SCD-Related TEAEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs were defined as AEs with onset on or after the date of informed consent until 28 days after last dose of study drug. Non-SCD-related TEAEs included all the PTs of TEAEs other than SCD- related TEAEs. The number of participants with any non-SCD-related TEAEs was reported in this outcome measure.
Time Frame: From date of informed consent up to 28 days after last dose of study drug (maximum up to 300.7 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
Participants | 59 | 49 | 52

3. Primary Outcome: Number of Participants With SCD-Related Treatment Emergent Serious Adverse Events (TESAEs)
Description: An SAE is an AE at any dose, in view of investigator resulted in any of following outcomes: death; life-threatening AE; inpatient hospitalization/prolongation of existing hospitalization; persistent/significant incapacity or disability; a congenital anomaly/birth defect and important medical events (IME) that may not result in death, be immediately life threatening; or require hospitalization may be considered serious when based upon medical judgement, they may jeopardize study participant and may require medical or surgical intervention to prevent one of outcomes listed in definition. TESAEs were defined as SAEs with onset on or after the date of informed consent until 28 days after last dose of study drug. Number of participants with SCD-Related TESAEs was reported in this outcome measure.
Time Frame: From date of informed consent up to 28 days after last dose of study drug (maximum up to 300.7 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
Participants | 39 | 33 | 22

4. Primary Outcome: Number of Participants With Non-SCD-Related TESAEs
Description: An SAE is an AE at any dose, in view of investigator resulted in any of following outcomes: death; life-threatening AE; inpatient hospitalization/prolongation of existing hospitalization; persistent/significant incapacity or disability; a congenital anomaly/birth defect and IME that may not result in death, be immediately life threatening; or require hospitalization may be considered serious when based upon medical judgement, they may jeopardize study participant and may require medical or surgical intervention to prevent one of outcomes listed in definition. TESAEs were defined as SAEs with onset on or after the date of informed consent until 28 days after last dose of study drug. Number of participants with non-SCD related TESAEs was reported in this outcome measure.
Time Frame: From date of informed consent up to 28 days after last dose of study drug (maximum up to 300.7 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
Participants | 18 | 14 | 15

5. Primary Outcome: Annualized Incidence Rate (Events Per Person Years) of SCD-Related Complications
Description: Annualized incidence rate was defined as total number of events (i.e. complications observed for all participants) divided by total person years. Total person-years= sum of participant summary period in years where summary period=date of informed consent until the earlier of 28 days after last dose of study drug or end of study date. SCD related complications included acute chest syndrome, cerebrovascular accident, hepatic sequestration, ocular icterus, osteonecrosis, pneumonia, priapism, pulmonary hypertension, retinopathy, sickle cell anaemia with crisis, skin ulcer and splenic sequestration. The 95% CI was based on exact Poisson confidence limits. Incidence rate of all SCD related complications is reported in this outcome measure.
Time Frame: From date of informed consent up to earlier of 28 days after last dose of study drug or end of study date (maximum up to 300.7 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per person years
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
Events per person years | 1.181 [1.031 to 1.347] | 1.084 [0.924 to 1.264] | 1.045 [0.905 to 1.200]

6. Primary Outcome: Annualized Incidence Rate (VOC Events Per Person Years) of On-Treatment Vaso-occlusive Crisis (VOCs)
Description: Annualized incidence rate was defined as total number of VOC events divided by total person years. Total person-years= sum of participant summary period in years where summary period=date of informed consent to last dose of study drug. VOC during the treatment period was defined as composite of acute painful crisis or acute chest syndrome (ACS) and included the following: moderate to severe pain lasting at least 2 hours; no explanation other than VOC; required oral or parenteral opioids, ketorolac, or other analgesics prescribed or directed by a healthcare professional. The 95% CI was based on exact Poisson confidence limits.
Time Frame: From date of informed consent to last dose of study drug (maximum up to 296.7 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: VOC events per person years
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 62 | 58 | 58
VOC events per person years | 1.038 [0.896 to 1.195] | 0.926 [0.778 to 1.095] | 0.889 [0.760 to 1.034]

7. Secondary Outcome: Change From Baseline in Hemoglobin Level at Week 48
Description: Change from baseline in hemoglobin at Week 48 was reported in this outcome measure. Baseline value was defined as the last available value (including Week 72, end of treatment [EOT], or end of study [EOS] visits in the parent study GBT440-031 [NCT03036813]) collected on or prior to first dose in GBT440-034.
Time Frame: Baseline, Week 48
Population: The safety population included all enrolled participants who received treatment with study drug voxelotor in the current study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Gram per deciliter (g/dL)
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 57 | 53 | 55
Gram per deciliter (g/dL)
  Baseline | 8.8 (1.32) | 9.0 (1.52) | 9.5 (1.61)
  Change at Week 48: number analyzed (Participants) | 40 | 35 | 39
  Change at Week 48 | 1.2 (1.50) | 0.7 (1.48) | 0.2 (1.15)

8. Secondary Outcome: Percent Change From Baseline in Reticulocytes Percentage at Week 48
Description: Percent change from baseline in reticulocytes percentage at Week 48 was reported in this outcome measure. Baseline value was defined as the last available value (including Week 72, EOT, or EOS visits in the parent study GBT440-031 [NCT03036813]) collected on or prior to first dose in GBT440-034.
Time Frame: Baseline, Week 48
Population: The safety population included all enrolled participants who received treatment with study drug voxelotor in the current study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 38 | 33 | 35
Percent change | -24.9 (58.13) | -15.3 (55.82) | -21.0 (81.29)

9. Secondary Outcome: Percent Change From Baseline in Absolute Reticulocytes at Week 48
Description: Percent change from baseline in absolute reticulocytes at Week 48 was reported in this outcome measure. Baseline value was defined as the last available value (including Week 72, EOT, or EOS visits in the parent study GBT440-031 [NCT03036813]) collected on or prior to first dose in GBT440-034.
Time Frame: Baseline, Week 48
Population: as for outcome 8
Measure: Median (Full Range); unit: Percent change
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 33 | 23 | 31
Percent change | -25.2 [-71.3 to 4123.7] | -25.7 [-76.4 to 139.2] | -25.8 [-74.9 to 259.6]

10. Secondary Outcome: Percent Change From Baseline in Indirect Bilirubin at Week 48
Description: Percent change from baseline in indirect bilirubin at Week 48 was reported in this outcome measure. Baseline value was defined as the last available value (including Week 72, EOT, or EOS visits in the parent study GBT440-031 [NCT03036813]) collected on or prior to first dose in GBT440-034.
Time Frame: Baseline, Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500 mg in GBT440-031(NCT03036813)
Number analyzed (Participants) | 35 | 32 | 33
Percent change | -39.3 (40.70) | 3.8 (70.47) | 1.2 (84.21)

ADVERSE EVENTS:
Time Frame: From date of informed consent up to 28 days after last dose of study drug (maximum up to 300.7 weeks)
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or one participant may have experienced both a serious and non-serious event during the study. Safety population included all enrolled participants who received treatment with study drug voxelotor in current study.
Groups:
- Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813): Participant who received voxelotor 900 mg in study GBT440-031 (NCT03036813) were administered voxelotor 1500 mg once daily in this study as long as they received clinical benefit and/or until the participant had access to voxelotor from an alternative source.
Arm/Group | Prior Treatment of Placebo in GBT440-031 (NCT03036813) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) | Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813)
All-Cause Mortality (participants affected / at risk) | 3/62 | 2/58 | 5/58
Serious Adverse Events (participants affected / at risk) | 42/62 | 35/58 | 26/58
Other Adverse Events (participants affected / at risk) | 60/62 | 50/58 | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Prior Treatment of Placebo in GBT440-031 (NCT03036813) (N=62) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) (N=58) | Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813) (N=58)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 36 | 32 | 20
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2
Gait disturbance (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 0 | 2
Osteomyelitis (Infections and infestations) | 3 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Coronavirus infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Malaria (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Parvovirus infection (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 1/34 | 1/23 | 2/21 — This adverse event was collected only in male participants.
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Prior Treatment of Placebo in GBT440-031 (NCT03036813) (N=62) | Prior Treatment of Voxelotor 900mg in GBT440-031(NCT03036813) (N=58) | Prior Treatment of Voxelotor 1500mg in GBT440-031(NCT03036813) (N=58)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 28 | 24 | 31
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2
Reticulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Microcytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Heart failure with reduced ejection fraction (Cardiac disorders) | 0 | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Retinopathy sickle cell (Eye disorders) | 1 | 1 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 2 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 2
Vitreous haemorrhage (Eye disorders) | 2 | 0 | 0
Astigmatism (Eye disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Retinal neovascularisation (Eye disorders) | 1 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 11 | 4
Vomiting (Gastrointestinal disorders) | 9 | 8 | 6
Diarrhoea (Gastrointestinal disorders) | 11 | 6 | 4
Constipation (Gastrointestinal disorders) | 5 | 9 | 5
Abdominal pain (Gastrointestinal disorders) | 8 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 6
Gastritis (Gastrointestinal disorders) | 1 | 2 | 5
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders) | 12 | 7 | 8
Pyrexia (General disorders) | 9 | 6 | 6
Fatigue (General disorders) | 5 | 5 | 5
Non-cardiac chest pain (General disorders) | 4 | 6 | 5
Oedema peripheral (General disorders) | 2 | 1 | 2
Influenza like illness (General disorders) | 1 | 0 | 3
Malaise (General disorders) | 1 | 2 | 1
Peripheral swelling (General disorders) | 1 | 1 | 1
Asthenia (General disorders) | 1 | 0 | 1
Administration site irritation (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Hernia pain (General disorders) | 1 | 0 | 0
Hunger (General disorders) | 0 | 1 | 0
Physical deconditioning (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0
Ocular icterus (Hepatobiliary disorders) | 3 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 4 | 14
COVID-19 (Infections and infestations) | 2 | 4 | 9
Nasopharyngitis (Infections and infestations) | 4 | 5 | 5
Urinary tract infection (Infections and infestations) | 5 | 6 | 3
Tonsillitis (Infections and infestations) | 6 | 1 | 6
Gastroenteritis (Infections and infestations) | 2 | 5 | 4
Malaria (Infections and infestations) | 2 | 5 | 3
Pneumonia (Infections and infestations) | 3 | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 2
Pharyngitis (Infections and infestations) | 2 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1 | 2
Infection (Infections and infestations) | 2 | 1 | 1
Influenza (Infections and infestations) | 1 | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 2 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Coronavirus infection (Infections and infestations) | 1 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Paraspinal abscess (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1
Penile infection (Infections and infestations) | 0 | 0 | 1
Pilonidal disease (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 0 | 1
Tinea capitis (Infections and infestations) | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract candidiasis (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vulval abscess (Infections and infestations) | 1 | 0 | 0
Wound sepsis (Infections and infestations) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 1 | 1
Cardiac murmur (Investigations) | 2 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood corticotrophin decreased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1
Foetal haemoglobin decreased (Investigations) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Helicobacter test positive (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Mean cell volume decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Pulmonary function test decreased (Investigations) | 0 | 0 | 1
Staphylococcus test positive (Investigations) | 0 | 0 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Haemochromatosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Multi-vitamin deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 9 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 9 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 16 | 10 | 14
Dizziness (Nervous system disorders) | 4 | 2 | 7
Lethargy (Nervous system disorders) | 2 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2 | 0
Migraine (Nervous system disorders) | 1 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Hemiparaesthesia (Nervous system disorders) | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1
Vestibular migraine (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Microalbuminuria (Renal and urinary disorders) | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal hypertrophy (Renal and urinary disorders) | 0 | 0 | 1
Renal injury (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Priapism (Reproductive system and breast disorders) | 3/34 | 3/23 | 4/21 — This adverse event was collected only in male participants.
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 3
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 2 | 0 | 0
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung hypoinflation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Menopause (Social circumstances) | 0 | 0 | 1
Hypotension (Vascular disorders) | 4 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0
Systolic hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT03573882/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT03573882/SAP_001.pdf